CLINICAL TRIAL: NCT07066436
Title: ImmunoMRI for Assessment of Tumor-associated Macrophages: A Prospective Study in Patients With Diffuse Large B-cell Lymphoma Receiving CAR T-cell or Bispecific Antibody Therapy
Brief Title: ImmunoMRI for Assessment of Tumor-associated Macrophages
Status: Not yet recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Marius Mayerhoefer, Professor, Principal Investigator, Medical University of Vienna
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: KLP5104424
Record Dates: First submitted 2025-06-24; First posted 2025-07-15 (Actual); Last update posted 2025-07-15 (Actual); Status verified 2025-07

CONDITIONS: DLBCL - Diffuse Large B Cell Lymphoma
MeSH Terms: conditions — Dendritic Cell Sarcoma, Interdigitating

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Intravenous injection of ferumoxytol as off-label MRI contrast agent for tracking of macrophages (Experimental): ImmunoMRI for tracking of TAMs will be integrated into 18F-FDG-PET/MRI scans that are performed for routine clinical purposes -i.e., assessment of disease extent before, and response assessment after/on treatment- to minimize patient discomfort and improve compliance.
  ImmunoMRI will be based on an iron sensitive fat-suppressed, fast spoiled gradient echo T2* mapping sequence, obtained before and after intravenous injection of the iron oxide nanoparticle ferumoxytol (commerical name: Feraheme).
  For each patient immunoMRI will be performed twice: before treatment, and 3-4 weeks after start of treatment (CAR T cells or bispecific antibodies).
  Interventions: Drug: MRI contrast-enhancing agents

INTERVENTIONS:
Drug: MRI contrast-enhancing agents — 1. Ferumoxytol will be injected as an off-label MRI contrast agent at a dose of 4 mg/kg body mass. For safety (in accordance with prior research), ferumoxytol will be diluted 1:4 in saline, and administered slowly over at least 15 minutes, with patient monitoring during and post injection.
  2. ImmunoMRI will be performed using an iron sensitive fat-suppressed, fast spoiled gradient echo T2* mapping sequence. At each time point (i.e. pre-treatment and post-treatment), T2* mapping will be performed before and ~24h after ferumoxytol injection.

SUMMARY:
About 35% of patients with a type of blood cancer called diffuse large B-cell lymphoma don't respond well to standard treatment or their cancer comes back. When this happens, newer treatments like CAR T-cell therapy (using modified immune cells) or bispecific antibodies (special proteins that help the immune system fight cancer) are an option. However, these treatments are only successful in about half the patients. It is currently difficult to predict which patients will respond to these treatments or experience serious side effects. This makes it hard to choose the best treatment plan for a given patient.

In this project, a special type of magnetic resonance imaging (MRI) scan will be used to track immune cells called macrophages that live around tumors. These cells can either help fight cancer or help cancer grow. By understanding how these cells behave, it may be possible to predict treatment success. The MRI technique involves injecting an iron-based substance called ferumoxytol, which can be used as an MRI contrast agent, into patients' veins. This contrast agent gets absorbed by the macrophages, making them visible on MRI scans throughout the entire body - not just one tumor spot. Sixty patients will be scanned before and after treatment (30 getting CAR T-cells, 30 getting bispecific antibodies), and results will be compared with tissue samples.

The goals are to predict which patients will go into complete remission, predict who will survive longer without cancer progression, and identify patients at risk for serious side effects like cytokine release syndrome. If successful, this imaging technique could help to personalize treatment choices, potentially improving outcomes while avoiding unnecessary toxicity in patients who will not benefit from these intensive therapies.

DETAILED DESCRIPTION:
Lymphomas are the most common types of blood cancer worldwide. Among these, diffuse large B-cell lymphoma (DLBCL) is both the most common overall and the most aggressive type, affecting about 4 out of every 100,000 people in Europe each year. This cancer typically causes noticeable symptoms and requires immediate treatment.

The World Health Organization recognizes several subtypes of DLBCL based on how the cancer cells look under a microscope, clinical features, and genetic characteristics. Some variants are particularly aggressive, especially those with multiple genetic abnormalities called "double-hit" or "triple-hit" lymphomas.

While many patients with DLBCL can be cured with intensive combination treatments that include both chemotherapy and immunotherapy, about 30-40% of patients experience cancer that comes back or does not respond to treatment. For these patients, traditional intensive treatments followed by stem cell transplants offer poor outcomes, with patients typically surviving only about 6 months. This urgent need has led researchers to develop new, more targeted therapeutic approaches, such as CAR T-cells and bispecific antibodies.

CAR T-Cell Therapy:

Reprogramming the Body's Own Defense System CAR T-cell therapy represents a groundbreaking approach to cancer treatment. This innovative treatment works by taking a patient's own immune cells (called T-cells) from their blood and genetically modifying them in a laboratory. These modified cells are programmed to specifically recognize and attack cancer cells. The process involves adding special receptors to the T-cells that can identify specific proteins on cancer cells, particularly one called CD19 that's commonly found on lymphoma cells. Once these engineered T-cells are infused back into the patient, they multiply and launch a targeted attack against the cancer. Currently, three CAR T-cell products are approved for clinical use, each with slightly different characteristics and side effect profiles. Major clinical trials have shown remarkable results, with complete remission rates of 65-66% compared to only 32-39% with standard treatments. Patients also experienced much longer periods without cancer progression. However, CAR T-cell therapy comes with significant challenges. The treatment can cause serious side effects in the majority of patients, including potentially life-threatening conditions called cytokine release syndrome (CRS) and immune effector cell-associated neurotoxicity syndrome (ICANS). Additionally, the treatment isn't immediately available because it requires collecting the patient's cells, modifying them in specialized facilities, and then manufacturing the personalized treatment-a process that can cause dangerous delays.

Bispecific Antibodies:

An Immediately Available Alternative Bispecific antibodies offer a promising alternative that's immediately available to patients. These engineered proteins work like molecular bridges, connecting the patient's existing T-cells directly to cancer cells. They target two different proteins simultaneously: CD3 on T-cells and CD20 on cancer cells.Two main bispecific antibodies, glofitamab and epcoritamab, have shown encouraging results in clinical studies. These treatments achieved response rates of 52-68% and complete remission rates of 39-57% in heavily pre-treated patients. Importantly, while these treatments can also cause CRS and ICANS, current data suggests these side effects are less common and less severe than with CAR T-cells.

The Hidden Players: Tumor-Associated Macrophages

Within every tumor, there's a complex ecosystem of different cell types, including immune cells called macrophages. These cells normally serve as the body's cleanup crew and help coordinate immune responses. However, in the tumor environment, these tumor-associated macrophages (TAMs) can behave in two very different ways. Some macrophages adopt an anti-tumor role (called M1 polarization), actively fighting against cancer cells and helping to present cancer proteins to other immune cells. However, others can become tumor-supporting (M2 polarization), actually helping tumors grow, spread, and resist treatment. The tumor-supporting M2 macrophages can suppress the very T-cells that CAR T-cell and bispecific antibody therapies depend on. They do this by depleting essential nutrients that T-cells need to function, producing anti-inflammatory substances that dampen immune responses, and directly blocking T-cell activation pathways. Understanding and measuring these TAMs could be crucial for predicting which patients will respond to these new treatments and which might experience serious side effects.

ImmunoMRI: A New Way to Make Macrophages Visible

Currently, physicians can only assess TAMs by taking small tissue samples (biopsies) from tumors. This approach has major limitations because it only examines a tiny fraction of the tumor and typically from just one location. Since cancer can vary significantly throughout the body, these small samples may not represent the full picture of what is happening with the immune system across all tumor sites. ImmunoMRI offers a revolutionary solution using a special type of MRI scan with an iron-based contrast agent called ferumoxytol. This agent is already FDA-approved for treating iron deficiency anemia, but it also has another unique property: it is taken up specifically by macrophages throughout the body. Patients receive an injection of ferumoxytol, and then 1-2 days later, they undergo a special MRI scan. The iron particles that have been absorbed by macrophages create distinctive changes in the MRI signal, allowing physicians to see and measure TAM levels throughout the entire body-not just in one small biopsy sample. This whole-body approach could provide a much more complete picture of the immune landscape across all tumor sites, potentially helping physicians better predict treatment responses and side effects.

Research Goals: Four Critical Questions

This research project, which will include sixty patients with relapsed/refratory DLBCL (30 treated with CAR T-cells, 30 treated with bispecific antibodies), aims to answer four important questions that could transform how physicians treat patients with this type of blood cancer:

Question 1: Does ImmunoMRI Accurately Reflect Macrophages in Lymphoma? The researchers will compare ImmunoMRI results with traditional tissue analysis to confirm that the imaging technique accurately reflects TAM levels. They will use special stains to identify different types of macrophages and determine whether the MRI technique better detects anti-tumor or tumor-supporting macrophages.

Working hypothesis: ImmunoMRI will show strong correlations with tissue analysis, particularly for the tumor-supporting M2-type macrophages that are expected to be more common in aggressive lymphomas.

Question 2: Are Changes in ImmunoMRI Related to Treatment Response? By comparing ImmunoMRI scans taken before and after treatment, researchers will determine if changes in TAM levels correlate with changes in tumor size and metabolic activity (measured by standard PET scans).

Working hypothesis: Treatments that successfully reduce TAM levels will also show corresponding decreases in tumor size and metabolic activity.

Question 3: Can ImmunoMRI Predict Long-term Outcomes? The study will test whether TAM levels measured before treatment, or how they change after treatment, can predict which patients will achieve complete remission or have better survival rates.

Working hypothesis: Patients with high TAM levels before treatment, or those whose TAM levels do not decrease much after treatment, will be more likely to have treatment-resistant cancer and shorter survival.

Question 4: Can ImmunoMRI Predict Dangerous Side Effects? Since macrophages play a key role in causing CRS and ICANS-the most serious side effects of these new treatments-researchers will explore whether ImmunoMRI can identify patients at higher risk for these complications.

Working hypothesis: Patients who develop CRS or ICANS will have higher TAM levels on their ImmunoMRI scans, either before or shortly after treatment.

Why This Research Matters

Currently, 50-60% of patients with relapsed or treatment-resistant DLBCL do not achieve lasting remission even with these revolutionary new treatments. Given the high cost and potential toxicity of CAR T-cell and bispecific antibody therapies, there is an urgent need for better ways to predict which patients will benefit and which might experience serious side effects.

ImmunoMRI could provide physicians with a new tool to:

1. Better select patients who are most likely to benefit from these expensive treatments
2. Predict and potentially prevent serious side effects
3. Monitor treatment response in real-time across the entire body
4. Develop more personalized treatment approaches

This research represents a significant step toward precision medicine in blood cancer treatment, potentially improving outcomes while reducing unnecessary toxicity and healthcare costs. By better understanding the complex interplay between cancer cells, immune cells, and these new treatments, physicians may be able to provide more effective, safer care for patients facing this challenging disease.

ELIGIBILITY:
Inclusion Criteria:

1. Pathology-proven relapsed/refractory DLBCL
2. Evidence of at least one anatomic site of tumor involvement on most recent prior imaging, e.g. CT, MRI, PET, or ultrasound, reflecting R/R DLBCL.
3. Ability to understand the study goals or outline and to give written informed consent.

Exclusion Criteria:

1. Clinically confirmed pregnancy for women, or breast-feeding women; for pre-menopausal women who do not use hormonal contraception, a pregnancy test with a negative result will be required.
2. Age below the specified minimum of 18 years.
3. Any type of anemia at baseline (due to potentially altered ferumoxytol uptake)
4. Impaired renal function / renal insufficiency
5. Known contraindication to MRI (per MRI Safety Guidelines, or conditions such as claustrophobia)
6. Known hypersensitivity to ferumoxytol or any of its components, or history of allergic reaction to any intravenous iron product.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-10 (Estimated); Primary Completion 2028-03 (Estimated); Study Completion 2028-09 (Estimated)

PRIMARY OUTCOMES:
Correlation between immunoMRI and M1 and M2 TAM-directed IHC | Through study completion, 3 years
  To determine the associations between pre-treatment immunoMRI metrics and IHC-based TAM levels, median/mean T2* will be calculated for each of the four IHC categories (score 1-4), separately for M1 and M2 TAMs, and Spearman rank correlation coefficients will be calculated.
Prediction of complete remission (CR) | Through study completion, 3 years
  Median/mean pre-treatment T2* and on-treatment T2* changes (relative to baseline), will be compared between patients achieving/not achieving complete remission (CR). Logistic regression analyses will be used to test combinations of pre-treatment T2* and △T2*, and respective SUV (standardized uptake values) and MTV (metabolic tumor volumes) on PET and VOL (morphologic volumes) on MRI
Prediction of 1-year overall survival (OS) | Through study completion, 3 years
  Median/mean pre-treatment T2* and on-treatment T2* changes (relative to baseline) will be compared between patients achieving/not achieving 1-year OS. Logistic regression analyses will be used to test combinations of pre-treatment T2* and △T2*, and respective SUV (standardized uptake values) and MTV (metabolic tumor volumes) on PET and VOL (morphologic volumes) on MRI, to predict 1-year OS.
Prediction of 1-year PFS | Through study completion, 3 years
  Median/mean pre-treatment T2* and on-treatment T2* changes (relative to baseline) will be compared between patients achieving/not achieving 1-year OS. Logistic regression analyses will be used to test combinations of pre-treatment T2* and △T2*, and respective SUV (standardized uptake values) and MTV (metabolic tumor volumes) on PET and VOL (morphologic volumes) on MRI, to predict 1-year OS.
Prediction of development of treatment toxicities (CRS, ICANS) | Through study completion, 3 years
  Median/mean pre-treatment T2*pre and on-treatment △T2* values will be compared between patients developing/not developing cytokine release syndrom (CRS) or immune effector cell-associated neurotoxicity syndrome (ICANS), and ROC analyses will be performed for each treatment group

SECONDARY OUTCOMES:
Correlation between post-treatment immunoMRI changes with changes in metabolic tumor activity and tumor size | Through study completion, 3 years
  To determine the association between early post-treatment changes in TAM levels and standard image-based tumor response, △T2* (post-treatment T2* - pretreatment T2*) will be correlated with respective △SUVs, △MTV, and △VOL, using Pearson and Spearman correlation coefficients, as appropriate.
Differences between males and females in terms of imaging metrics | Through study completion, 3 years
  Comparison of T2* values between males and females
Differences between males and females in terms of IHC scores | Through study completion, 3 years
  Comparison of TAM IHC scores between males and females
Differences between males and females in terms of treatment response | Through study completion, 3 years
  Comparison of percentages of males and females achieving complete remission (CR)
Differences between males and females in terms of 1-year OS | Through study completion, 3 years
  Comparison of percentages of males and females achieving 1-year overall survival (OS)
Differences between males and females in terms of 1-year PFS | Through study completion, 3 years
  Comparison of percentages of males and females achieving 1-year progression-free survival (PFS)

CONTACTS AND LOCATIONS:
Overall Officials: Marius E Mayerhoefer, MD, PhD, Principal Investigator — Medical University of Vienna
Locations (1):
- Medical University of Vienna, Vienna, Vienna, Austria

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Neelapu SS, Tummala S, Kebriaei P, Wierda W, Gutierrez C, Locke FL, Komanduri KV, Lin Y, Jain N, Daver N, Westin J, Gulbis AM, Loghin ME, de Groot JF, Adkins S, Davis SE, Rezvani K, Hwu P, Shpall EJ. Chimeric antigen receptor T-cell therapy - assessment and management of toxicities. Nat Rev Clin Oncol. 2018 Jan;15(1):47-62. doi: 10.1038/nrclinonc.2017.148. Epub 2017 Sep 19. PMID 28925994
- [Background] Kamdar M, Solomon SR, Arnason J, Johnston PB, Glass B, Bachanova V, Ibrahimi S, Mielke S, Mutsaers P, Hernandez-Ilizaliturri F, Izutsu K, Morschhauser F, Lunning M, Maloney DG, Crotta A, Montheard S, Previtali A, Stepan L, Ogasawara K, Mack T, Abramson JS; TRANSFORM Investigators. Lisocabtagene maraleucel versus standard of care with salvage chemotherapy followed by autologous stem cell transplantation as second-line treatment in patients with relapsed or refractory large B-cell lymphoma (TRANSFORM): results from an interim analysis of an open-label, randomised, phase 3 trial. Lancet. 2022 Jun 18;399(10343):2294-2308. doi: 10.1016/S0140-6736(22)00662-6. PMID 35717989
- [Background] Kochenderfer JN, Dudley ME, Kassim SH, Somerville RP, Carpenter RO, Stetler-Stevenson M, Yang JC, Phan GQ, Hughes MS, Sherry RM, Raffeld M, Feldman S, Lu L, Li YF, Ngo LT, Goy A, Feldman T, Spaner DE, Wang ML, Chen CC, Kranick SM, Nath A, Nathan DA, Morton KE, Toomey MA, Rosenberg SA. Chemotherapy-refractory diffuse large B-cell lymphoma and indolent B-cell malignancies can be effectively treated with autologous T cells expressing an anti-CD19 chimeric antigen receptor. J Clin Oncol. 2015 Feb 20;33(6):540-9. doi: 10.1200/JCO.2014.56.2025. Epub 2014 Aug 25. PMID 25154820
- [Background] Nguyen KL, Yoshida T, Kathuria-Prakash N, Zaki IH, Varallyay CG, Semple SI, Saouaf R, Rigsby CK, Stoumpos S, Whitehead KK, Griffin LM, Saloner D, Hope MD, Prince MR, Fogel MA, Schiebler ML, Roditi GH, Radjenovic A, Newby DE, Neuwelt EA, Bashir MR, Hu P, Finn JP. Multicenter Safety and Practice for Off-Label Diagnostic Use of Ferumoxytol in MRI. Radiology. 2019 Dec;293(3):554-564. doi: 10.1148/radiol.2019190477. Epub 2019 Oct 22. PMID 31638489
- [Background] Aghighi M, Theruvath AJ, Pareek A, Pisani LL, Alford R, Muehe AM, Sethi TK, Holdsworth SJ, Hazard FK, Gratzinger D, Luna-Fineman S, Advani R, Spunt SL, Daldrup-Link HE. Magnetic Resonance Imaging of Tumor-Associated Macrophages: Clinical Translation. Clin Cancer Res. 2018 Sep 1;24(17):4110-4118. doi: 10.1158/1078-0432.CCR-18-0673. Epub 2018 May 15. PMID 29764855